CLINICAL TRIAL: NCT06395675
Title: Clinical Evaluation of the ID NOW™ CT/NG Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Abbott Diagnostics Scarborough
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Chlamydia Trachomatis Infection; Neisseria Gonorrheae Infection; Asymptomatic Condition
MeSH Terms: conditions — Gonorrhea; Asymptomatic Diseases

STUDY DESIGN:
Intervention Model Description: Each female participant will provide a 20-50 mL first-catch urine (FCU) sample, one (1) self-collected vaginal swab sample (SVS) and three (3) clinician-collected vaginal swabs (CVS). Each male participant will provide a 20-50 mL first-catch urine sample. Standard of care (SOC) samples should be collected first prior to clinical trial specimen collection If sites use urine as SOC, then SOC urine sample can be taken from the untreated sterile urine cup provided to collect first catch urine for this study. Samples will be collected, handled, stored, shipped, and tested according to the applicable package insert(s), as appropriate. The site will record the order of sample collection for each participant. The remaining urine will be aliquoted into applicable transport.
  tubes for each comparator method (3 tubes) and one (1) retained urine sample (5mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Female/Male collection (Experimental): Each female participant will provide a 20-50 mL first-catch urine sample, and one (1) self-collected vaginal swab sample and three (3) clinician-collected vaginal swabs. Each male participant will provide a 20-50 mL first-catch urine sample.
  Each urine sample will be collected in an untreated sterile urine cup. The site staff will test 1.5 ml of urine directly from the specimen cup with ID NOW within two (2) hours of collection. The remaining urine will be aliquoted into applicable transport tubes for each comparator.
  One (1) self-collected vaginal swab will be collected by the participant in a clinical setting and tested on the device within 2 hours. Three (3) vaginal swabs will be collected by the clinician according to institutional procedures and manufacturer's instructions, one for each of the three (3) NAATs for comparator testing. For comparator tests, the order of CVS sample collection will be randomized.
  Interventions: Diagnostic Test: ID NOW™

INTERVENTIONS:
Diagnostic Test: ID NOW™ — The ID NOW™ CT/NG is an in vitro qualitative molecular assay for the rapid differential.
  detection of Chlamydia trachomatis (CT) and Neisseria gonorrhoeae (NG) in urine, and self-collected vaginal swabs (SVS) in symptomatic and asymptomatic individuals.

SUMMARY:
The objective of this study is to determine the performance of the ID NOW™ CT/NG test in male urine, female urine, and self-collected vaginal swabs when tested by intended users (i.e., untrained operators). ID NOW™ CT/NG test results will be compared to results from up to three (3) FDA cleared CT/NG nucleic acid amplification tests (NAATs) for each sample type.

DETAILED DESCRIPTION:
This is a global study and will be conducted at approximately thirty (30) US clinical study sites and up to five (5) study sites OUS in Europe, UK and Africa. The participating sites in the US will be in different geographical areas. Up to 30% of NG positive female participants (by composite Comparative Result (CCR)) may participate from OUS sites. ID NOW™ testing will be conducted by untrained operators (i.e., site staff with limited or no training or hands-on experience in conducting laboratory testing).

Approximately 7,100 participants will be enrolled. Consented participants will provide samples for ID NOW™ CT/NG and comparator assay testing. Each female participant will provide a 20-50 mL first-catch urine (FCU) sample, one (1) self-collected vaginal swab sample (SVS) and three (3) clinician-collected vaginal swabs (CVS). Each male participant will provide a 20-50 mL first-catch urine sample. Standard of care (SOC) samples should be collected first prior to clinical trial specimen collection. SOC vaginal swab should be collected before vaginal swabs (self- and clinician-collected) are collected as part of the study. If sites use urine as SOC, then SOC urine sample can be taken from the untreated sterile urine cup provided to collect first catch urine for this study.

Samples will be collected, handled, stored, shipped, and tested according to the applicable Package Insert(s), as appropriate. The site will record the order of sample collection for each participant. ID NOW™ CT/NG testing will be conducted on fresh samples. The sites will ship samples to a central laboratory for testing with up to three (3) FDA cleared CT/NG nucleic acid amplification tests (NAATs) according to the appropriate package insert(s). The central laboratory may be located outside of the clinical site(s) country for OUS sites and thus require shipping of samples outside of the clinical sites(s) country as per compliance.

Each urine sample will be collected in an untreated sterile urine cup provided by Sponsor. The site staff will ensure the urine cup is capped and then invert the urine cup five (5) times to mix. Once inverted five (5) times, site staff will test 1.5 ml of urine directly from the specimen cup with ID NOW™ CT/NG within two (2) hours of collection. The remaining urine will be aliquoted into applicable transport tubes for each comparator method (3 tubes) and one (1) retained urine sample (5mL). One (1) self-collected vaginal swab will be collected and placed in Sample Elution buffer by the participant in a private clinical setting. The participant will be provided with instructions on appropriate collection. Three (3) additional vaginal swabs will be collected by a clinician for each of the three (3) comparator tests per Product Inserts. The order in which SVS and CVS are collected will be randomized by Participant ID number. For participants with an odd-numbered Participant ID, the SVS will be collected first, followed by the three (3) CVS. For participants with an even-numbered Participant ID, the three (3) CVS will be collected first, followed by the SVS. For comparator tests, the order of CVS sample collection will be randomized (Appendix B). A portion (1.5 ml) of SVS in buffer will be tested with the ID NOW™ CT/NG test within 2 hours of sample collection. ID NOW™ CT/NG test results are investigational and will not be used for patient diagnosis or to guide treatment. After ID NOW™ CT/NG testing, leftover vaginal swab eluate and urine samples will be stored at the site according to Sponsor instructions and in the case that further testing is needed, shipped to an Abbott location/central laboratory at the Sponsor's request. No personally identifiable testing for human DNA will be performed on any samples obtained from this study. The Abbott location or central laboratory may be located outside of the clinical site(s) country for OUS sites and thus require shipping of samples outside of the clinical sites(s) country.

The Sponsor will perform data analysis. The results of the ID NOW™ CT/NG test will be presented separately for CT and NG. ID NOW™ CT/NG test results will be presented by sample type, by sex, and by symptomatic and asymptomatic status. POC Link functionality may be established with each ID NOW™ Instrument for remote connectivity.

ELIGIBILITY:
Inclusion Criteria: Participants providing vaginal samples and urine

* Aged 14 years or older in US or 18 years or older in OUS
* Sexual activity within the past six (6) months
* Asymptomatic and presenting for STI screening, OR Symptomatic with suspected sexually transmitted infection and one or more of the following symptoms:
* lower abdominal, pelvic, or adnexal pain
* abnormal vaginal discharge
* pain or discomfort with sexual intercourse
* bleeding between menstrual cycles and/or after sex
* pain, discomfort, frequency, or urgency with urination
* Able and willing to provide approximately 20-50 mL first-catch urine sample, one (1) self-collected vaginal swab, and three (3) Clinician-collected vaginal swabs.
* The participant and/or legally authorized representative is willing to undergo the informed consent process prior to study participation (a minor will need the documented assent and consent of their parent or legal guardian, unless the site has an IRB/EC (Institutional Review Board/Ethics Committee) approved waiver for parental consent for minors)

Inclusion Criteria -Participants providing urine only

* Aged 14 years or older in US or 18 years or older in OUS
* Sexual activity within the past six (6) months
* Asymptomatic and presenting for STI screening, OR
* Symptomatic with suspected sexually transmitted infection and one or more of the following symptoms:
* discharge from penis
* burning sensation during urination
* pain or swelling in one or both testicles
* Able and willing to provide approximately 20-50 mL first-catch urine sample
* The participant and/or legally authorized representative is willing to undergo the informed consent process prior to study participation (a minor will need the documented assent and consent of their parent or legal guardian, unless the site has an IRB/EC approved waiver for parental consent for minors)

Exclusion Criteria: All participants

* Reported using or having completed antimicrobial therapy within 14 days of enrollment in the study
* Urination within the previous one (1) hour
* Unable to meet all inclusion criteria as listed
* Already participated in the study

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7100 (Estimated)
Dates: Start 2024-07-09 (Estimated); Primary Completion 2025-01-09 (Estimated); Study Completion 2025-01-09 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the positive percent agreement (PPA) and negative percent agreement (NPA) | "up to 24 months"
  The primary objective of this study is to demonstrate the positive percent agreement (PPA) and negative percent agreement (NPA) of the ID NOW™ CT/NG test using first catch urine tested directly, and self-collected vaginal swabs (SVS) placed in Sample Elution buffer immediately after collection.
  ID NOW™ CT/NG test results will be compared to results from up to three (3) FDA cleared CT/NG nucleic acid amplification tests (NAATs) for each sample type.

SECONDARY OUTCOMES:
Demonstrate the accuracy of the ID NOW™ CT/NG test in the hands of untrained users by a usability questionnaire. | "up to 24 months"
  The secondary objective of this study is to demonstrate the accuracy of the ID NOW™ CT/NG test in the hands of untrained users, which are "intended users" in a point of care (POC) Clinical Laboratory Improvement Amendments of 1988 (CLIA) moderate, high or waived complexity test environment.
  Each test operator will be given a user evaluation questionnaire once to assess the usability of the device.

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Crescent Care Sexual Health Clinic, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No